CLINICAL TRIAL: NCT04349566
Title: Fast Troponin as a Biomarker to Assess Exercise-induced Muscle Damage in Muscle Diseases
Status: Completed | Type: Observational
Sponsor: Mads Peter Godtfeldt Stemmerik (Other)
Collaborators: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mads Peter Godtfeldt Stemmerik, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: FAST TROPONIN
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Becker Muscular Dystrophy; McArdle Disease; Limb-Girdle Muscular Dystrophy Type 2
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Glycogen Storage Disease Type V; Limb-girdle muscular dystrophy type 2A

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to explore the biomarker Fast Troponins response to exercise in patients with Becker muscular dystrophy, Limb-girdle muscular dystrophy and McArdle disease

ELIGIBILITY:
Inclusion Criteria:

* The ability to cycle
* No concurrent medical condition that could interfere with interpretation of the results
* Molecular diagnosis of the specific condition in specified patient groups or healthy control
* No active muscle injury on the test day (caused by recent exercise, seizures, trauma, etc.)

Exclusion Criteria:

* Competing conditions at risk of compromising the results of the study
* Cardiac or pulmonary disease contraindicating peak exercise testing or strenuous exercise
* Veins that are too difficult to puncture for blood sampling, evaluated by the investigator
* Severe muscle weakness, that prevents the subject completing the exercise test, evaluated by the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with McArdle disease and patients with two sub-typesof Limb-girdle and Becker muscular dystrophies will be included as well as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers | 24 hours
  Change in Fast and slow Troponin I after muscle damage

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Research Unit, 3342, Copenhagen, Denmark